CLINICAL TRIAL: NCT03631316
Title: Comparison on Pharmacokinetic Parameters of Innovative Valganciclovir Versus Generic Valganciclovir in Kidney Transplant Recipients
Brief Title: Pharmacokinetic Parameters of Innovative Valganciclovir Versus Generic Valganciclovir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luis Eduardo Morales Buenrostro (Other)
Responsible Party: Sponsor-Investigator, Luis Eduardo Morales Buenrostro, Clinical Professor of Nephrology, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Organization: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2260
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Kidney Transplantation; Cytomegalovirus Infections; Pharmacokinetics; Therapeutic Equivalency
Keywords: valganciclovir; kidney transplantation; pharmacokinetics
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

STUDY DESIGN:
Intervention Model Description: Pharmacovigilance study, prospective, observational, analytical, single center, cross over design, with random assignment to the sequence of both formulations in the same patient. Our aim will be compare the pharmacokinetic parameters of the innovative versus generic formulation of valGCV in renal transplant recipients under valGCV prophylaxis in the early posttransplant stage.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each participant will take both formulations. Groups will be formed regarding the order in which the different formulations of valganciclovir will be analyzed. Both formulations will be given in two identical container numbered in the specific order assigned. The order of administration of the drug will be randomized, neither the researcher nor the patient will know the order of the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generic valganciclovir (Experimental): Participants will receive generic formulation (Pisa) of valganciclovir, 450 mg tablets, total dosage 900 mg daily for 4 days.
  Interventions: Drug: Generic Valganciclovir
- Innovative valganciclovir (Active Comparator): The same participant will receive innovative drug valcyte (roche), 450 mg tablets, total dosage 900 mg daily during 4 days.
  Interventions: Drug: Innovative Valganciclovir

INTERVENTIONS:
Drug: Generic Valganciclovir — 900 mg daily during 4 days
  Other Names: Valganciclovir Pisa
  Arms: Generic valganciclovir
Drug: Innovative Valganciclovir — 900 mg daily during 4 days
  Other Names: Valcyte
  Arms: Innovative valganciclovir

SUMMARY:
Cytomegalovirus (CMV) is the most common opportunistic viral pathogen in solid organ transplant receptors (SOTR). In Mexico, the experience using generic immunosuppressants have been demonstrated a wide variation in the pharmacokinetic parameters between generic and innovative formulation, resulting in a suboptimal absorption of the drug and reaching infratherapeutic trough levels in blood. In this study the investigators will compare the pharmacokinetic parameters of innovative and generic valganciclovir in renal transplant recipients.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is the most common opportunistic viral pathogen in solid organ transplant receptors (SOTR). In the absence of prophylaxis, the frequency of CMV disease in high-risk recipients (R- / D +) is 60% and 20% for intermediate-risk patients (R + / D + or -). For universal prophylaxis, the antivirals most commonly used are valganciclovir (valGCV) and IV ganciclovir. ValGCV, a prodrug of ganciclovir, has a bioavailability of 60%, which represents more than 10 times that those obtained with ganciclovir.

Pharmacokinetic studies of Valganciclovir in SOTR have been demonstrated that insufficient doses can diminish its clinical efficacy and the development of viral resistance, while excessive doses can increase its toxicity.

The risk of viremia may be associated with ineffective plasma doses, as described by Wiltshire et al., where values of the area under the curve (AUC) between 40 and 50 μg/h/ml were associated with a lower incidence of viremia, while lower AUC values are associated with an increase 8 times more for viral replication rates. As a result, pharmacokinetic studies in SOTR guide the investigators in continuing with the research of their clinical impact.

A generic drug before their release to the market needs to show that is bioequivalent with the innovative drug, assuming that it has the same therapeutic effects.

The studies for demonstrate bioequivalence are carried out in controlled conditions with healthy participants, different of SOTR characteristics as: age, gender, race, comorbidities and concomitant medication. In addition, the excipients used in generic drug are different from those of the innovative drug, so the properties of the formulation can be modified (particle size or half-life), therefore, the efficacy and drug safety.

The primary outcome will be compare the pharmacokinetic parameters of the innovative versus generic formulation of valGCV in renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form for the study
* Age between 18 and 70 years
* Kidney transplant recipients who are stable during their follow-up
* Kidney transplant recipients between day 31 and 90 post-transplant surgery
* Kidney transplant recipients under prophylaxis with valganciclovir

Exclusion Criteria:

* Participants who can not stay 12 hours at the hospital for taking the blood samples.
* Participants with an acute rejection event
* Participants with active cytomegalovirus disease
* Participants with measurements of pharmacokinetic parameters with a single formulation without comparator
* Participants that withdraw their informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve, AUC (ng/h/mL) | At day 4 of treatment
  AUC (ngh/mL) in both drugs (innovative and generic)

SECONDARY OUTCOMES:
Maximum serum concentration, Cmax (ng/mL) | At day 4 of treatment
  Cmax (ng/mL) in both drugs (innovative and generic)
Initial concentration, C0 (ng/mL) | At day 4 of treatment
  C0 (ng/mL) in both drugs (innovative and generic)
Total clearance of the drug, CL/F (L/h) | At day 4 of treatment
  CL/F (L/h), in both drugs (innovative and generic)
Distribution volume, Vd/F (L/h) | At day 4 of treatment
  Vd/F (L/h), in both drugs (innovative and generic)

CONTACTS AND LOCATIONS:
Overall Officials: Luis E Morales-Buenrostro, PhD, Principal Investigator — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No